CLINICAL TRIAL: NCT02600325
Title: Grazoprevir (MK-5172)+ Elbasvir (MK-8742) for the Treatment of Acute Hepatitis C Genotype 1/4. The Dutch Acute HCV in HIV Study (DAHHS-2)
Brief Title: Dutch Acute HCV in HIV Study (DAHHS-2): Grazoprevir/Elbasvir for Acute HCV
Acronym: DAHHS-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Bart Rijnders, Dr., Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL2015-003210-24
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Results first posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-04

CONDITIONS: Acute Hepatitis C; Human Immunodeficiency Virus; Hepatitis C
Keywords: Acute Hepatitis C; Human Immunodeficiency virus; Grazoprevir; Elbasvir
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C | interventions — grazoprevir; elbasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Grazoprevir/elbasvir single tablet regimen (100/50mg)
  Interventions: Drug: Grazoprevir/Elbasvir 100mg/50mg

INTERVENTIONS:
Drug: Grazoprevir/Elbasvir 100mg/50mg — Grazoprevir/Elbasvir 100mg/50mg

SUMMARY:
New and recently EMA/FDA approved direct acting antiviral (DAA) combination therapies cure 95% or more of the patients chronically infected with HCV genotype 1 and 4. Grazoprevir (MK-5172) and elbasvir (MK-8742) combination therapy is such a, albeit not yet EMA/FDA approved combination DAA therapy.

It is likely that the synergistic effect of the host's immune response and antiviral therapy when given during the first 6 months of HCV infection makes antiviral therapy during acute HCV infection more effective. In this study the investigators would like to document that treatment of acute HCV with grazoprevir (MK-5172), elbasvir (MK-8742) is effective and can ben shortened from 12 to 8 weeks for HCV genotype 1 and 4 infection without substantial loss in efficacy.

Study design and intervention:

Prospective open label interventional clinical trial in which 80 acute HCV genotype 1 or 4 patients co-infected with HIV will receive 8 weeks of grazoprevir and elbasvir (a once-daily combination tablet).

Study population:

80 Adult HIV positive patients with an acute HCV genotype 1 or 4 infection from 10 HIV treatment centers in the Netherlands and Belgium will be included.

Primary endpoint: Sustained viral response (SVR) 12 weeks after the end of therapy in ITT study population (=genotype 1 and 4).

DETAILED DESCRIPTION:
Rationale:

Over the last 2 years, the treatment of chronic HCV underwent an enormous change in a positive way. New and recently EMA approved direct acting antiviral (DAA) combination therapies cure as 95% or more of the patients chronically infected with HCV genotype 1 and 4. Grazoprevir (MK-5172) and elbasvir (MK-8742) combination therapy is such a combination DAA therapy. Two recent phase II and 1 phase III clinical trial showed that chronic HCV genotype 1 can be cured with 12 weeks of combination therapy with grazoprevir and elabsvir with a 97% cure in HIV-HCV co-infected patients in the phase III C-Edge co-infection study. However, none of these new HCV therapies have been well studied for the treatment of acute HCV and are therefore not registered for this indication. The only treatment approved for acute HCV is interferon. Interferon based therapy for the treatment of HCV has been shown to be much more effective when given during the acute phase of the HCV infection than at a time when the infection has become chronic. A likely explanation for this difference in success for acute versus chronic HCV therapy is a substantial immune response that is present during the acute phase of HCV infection, but becomes exhausted during chronic infection. This potent immune response is broadly targeted against various HCV epitopes and eradicates approximately 20% of HCV infections within the first 12 to 18 months of infection. However, spontaneous cure of HCV becomes very rare after the first 12 to 18 months of infection due to immune exhaustion. It is likely that the synergistic effect of the host's immune response and antiviral therapy when given during the first 6 months of HCV infection makes direct acting antiviral therapy during acute HCV infection more effective.

Objectives:

To document that treatment of acute HCV with grazoprevir (MK-5172), elbasvir (MK-8742) is effective. To show that, due to the host's immune response at the time of an acute HCV infection, the duration of therapy with grazoprevir (MK-5172) and elbasvir (MK-8742) for acute HCV genotype 1 and 4 infections can be shortened from 12 to 8 weeks without substantial loss in efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. HIV positive
2. Acute HCV genotype 1 or 4 infection (≤26 weeks old at the baseline visit)

Exclusion Criteria:

1. Not on cART and a CD4 <500 at the time of screening
2. Patients on cART for >6 months with a HIV viral load >400 copies
3. Disallowed co-medication that cannot be stopped or replaced
4. History of liver cirrhosis of any etiology. Inclusion of patients with a chronic well-controlled HBV (HBV-DNA <below the limit of detection) is allowed if fibroscan excludes >F1 fibrosis
5. Protease inhibitor based and NNRTI based cART regimens are not allowed. Therefore, the inability to switch to a HAART regimen consisting of 2 nucleoside/tide reverse transcriptase inhibitors and an allowed third agent which can be raltegravir (Isentress®) 400mg BID, dolutegravir (Tivicay) 50mg QD or rilpivirine 25mg QD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: B Rijnders, PhD, Principal Investigator — Erasmus Medical Center
Locations (9):
- Institute of Tropical Medicine Antwerp (ITG), Antwerp, Belgium
- Netherlands (8):
  - Erasmus Medical Center (EMC), Rotterdam, South Holland
  - Onze Lieve Vrouwe Gasthuis (OLVG), Amsterdam
  - Slotervaart Hospital, Amsterdam
  - Rijnstate Hospital, Arnhem
  - University Medical Center Groningen (UMCG), Groningen
  - Maastricht University Medical Center (MUMC), Maastricht
  - Radbout University Medical Center, Nijmegen
  - Utrecht Medical University Center (UMCU), Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Popping S, Cuypers L, Claassen MAA, van den Berk GE, De Weggheleire A, Arends JE, Boerekamps A, Molenkamp R, Koopmans MPG, Verbon A, Boucher CAB, Rijnders B, van de Vijver DAMC. Persistent Transmission of HCV among Men Who Have Sex with Men despite Widespread Screening and Treatment with Direct-Acting Antivirals. Viruses. 2022 Sep 2;14(9):1953. doi: 10.3390/v14091953. PMID 36146760
- [Derived] Boerekamps A, De Weggheleire A, van den Berk GE, Lauw FN, Claassen MAA, Posthouwer D, Bierman WF, Hullegie SJ, Popping S, van de Vijver DACM, Dofferhoff ASM, Kootstra GJ, Leyten EM, den Hollander J, van Kasteren ME, Soetekouw R, Ammerlaan HSM, Schinkel J, Florence E, Arends JE, Rijnders BJA. Treatment of acute hepatitis C genotypes 1 and 4 with 8 weeks of grazoprevir plus elbasvir (DAHHS2): an open-label, multicentre, single-arm, phase 3b trial. Lancet Gastroenterol Hepatol. 2019 Apr;4(4):269-277. doi: 10.1016/S2468-1253(18)30414-X. Epub 2019 Jan 17. PMID 30660617

RESULTS

PARTICIPANT FLOW:
Groups:
- Grazoprevir/Elbasvir 100mg/50mg: Grazoprevir/elbasvir single tablet regimen (100/50mg)
  Grazoprevir/Elbasvir 100mg/50mg: Grazoprevir/Elbasvir 100mg/50mg
Period: Overall Study
Arm/Group | Grazoprevir/Elbasvir 100mg/50mg
Started | 80
Completed | 80
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: G/E 8 weeks
Arm/Group | Treatment Arm
Number analyzed (Participants) | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 80
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 72
  More than one race | 0
  Unknown or Not Reported | 8

OUTCOME MEASURES:

1. Primary Outcome: SVR12 (Reinfection Not Considered Failure)
Description: Sustained viral response (SVR) 12 weeks after the end of therapy in all patients who started treatment in which reinfections are not considered failure
Time Frame: 12 weeks
Measure: Number; unit: participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 80
participants | 79

2. Secondary Outcome: SVR12 (Reinfection Equals Failure)
Description: Sustained viral response (SVR) 12 weeks after the end of therapy in all patients who started treatment in which reinfections are considered failure
Time Frame: week 12
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 80
Participants | 75

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 2/80
Other Adverse Events (participants affected / at risk) | 43/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=80)
traumatic rectal bleeding (Gastrointestinal disorders) | 1 (1) — Unrelated SAE
Elective low back surgery (Musculoskeletal and connective tissue disorders) | 1 (1) — Unrelated SAE
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=80)
Fatique (General disorders) | 11 (11)
headache (General disorders) | 7 (7)
insomnia (General disorders) | 7 (7)
mood changes (General disorders) | 5 (5)
dyspepsia (Gastrointestinal disorders) | 5 (5)
concentration impairment (General disorders) | 4 (4)
dizziness (General disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/25/NCT02600325/Prot_SAP_000.pdf